CLINICAL TRIAL: NCT00324311
Title: Enzymatic Debridement in Burns Patients (Children & Adults): A Comparison to Standard of Care (Protocol MW 2004-11-02)
Brief Title: Enzymatic Debridement in Burns Patients: A Comparison to Standard of Care
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MediWound Ltd (Industry)
Responsible Party: Siyu Liu, Vice President, North American Innovative Research & Development and Head of Global Clinical Operations ), Teva Neuroscience
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MW2004-11-02
Record Dates: First submitted 2006-05-10; First posted 2006-05-11 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2009-07

CONDITIONS: Burn
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DGD (Experimental)
  Interventions: Drug: DGD
- SOC (Active Comparator)
  Interventions: Drug: DGD

INTERVENTIONS:
Drug: DGD — Lyophilized, sterile mixture of proteolyzed enzymes; mixed with gel,for topical application.

SUMMARY:
Burns represent one of the most severe and dreaded traumas. Burned and traumatized tissue is known as eschar. The dead eschar, if not removed, often becomes heavily contaminated and is the source of local and/or systemic infection or sepsis. The local inflammation and infection destroy healthy surrounding tissues and extends the original damage. In order to prevent these complications, and in order to minimize the risk of infection, it is imperative to evaluate the burn and remove all of the offending eschar at the earliest possible opportunity. This removal of dead tissue is termed "debridement".

The most direct debridement method for eschar removal is surgery. Traditional, conservative non-surgical debridement is a lengthy process which often involves many complications.

The objective of this study is to evaluate the safety and enzymatic debriding efficacy of Debrase Gel Dressing (DGD) in hospitalized patients with deep partial thickness and/or full thickness thermal burns and to compare DGD to standard of care (SOC).

DETAILED DESCRIPTION:
Completed study.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 4 years to 55 years of age,
2. Thermal burns caused by fire/flame, scalds or contact,
3. Deep partial thickness (mixed deep dermal) and/or full thickness (3°) burn wounds ≥ 5% and ≤ 30% Total Body Surface Area (TBSA); all these wounds must receive study treatment,
4. At least one wound of ≥ 2% TBSA deep partial thickness and/or full thickness burn,
5. Total burn wounds ≤ 30% TBSA,
6. Signed written informed consent.

Exclusion Criteria:

1. Deep partial thickness and/or full thickness facial burn wounds, > 0.5% TBSA; study treatment of facial burns is not allowed,
2. Study treatment of perineal and/or genital burns (A patient with these wounds may be enrolled but the wounds may not be designated as target wounds),
3. Circumferential anterior/posterior trunk full thickness fire/flame burns, > 15% TBSA, (Circumferential is defined as encircling ≥ 80% of the trunk circumference.)
4. Pre-enrollment escharotomy,
5. Heavily contaminated burns or pre-existing infections,
6. Signs that may indicate smoke inhalation,
7. General condition of patient would contraindicate surgery,
8. Pregnant women (positive pregnancy test) or nursing mothers,
9. Poorly controlled diabetes mellitus (HbA1c>9%),
10. Cardio-pulmonary disease (MI within 4 weeks prior to injury, pulmonary hypertension, COPD or pre-existing oxygen-dependent pulmonary diseases),
11. Pre-existing diseases which interfere with circulation (PVD, edema, lymphedema, surgery to the regional lymph nodes, obesity, varicose veins),
12. Immediate life threatening conditions (such as immuno-compromising diseases, life threatening trauma, severe pre-existing coagulation disorder, cardiovascular, liver or neoplastic disease),

Ages: 4 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 182 (Actual)
Dates: Start 2005-12; Primary Completion 2009-10 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Co-primary: % treated wound excised (by tangential/minor/Versajet excision) or dermabrasion, in first surgery, of deep partial wounds | Surgical excision/dermabrasion performed as initial debridement (surgical SOC group) or as first post-debridement procedure (DGD or non-surgical SOC groups)
Co-primary: % treated wound autografted of deep partial wounds | Post-debridement autografts

SECONDARY OUTCOMES:
% treated wound excised (by tangential/minor/Versajet excision) or dermabrasion, in first surgery, for all wounds | As for primary endpoint
Time to complete wound closure | % epithelialization assessed post-debridement at weekly intervals until all a patient's wounds closed
Timely eschar removal | Debridement procedures
Blood loss | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Lior Rosenberg, MD, Study Chair — MediWound Ltd
Locations (17):
- Royal Hospital Perth, Perth, Western Australia, Australia
- Brazil (2):
  - Pronto Socorro para Queimaduras de Goiania, Goiânia
  - Hospital do Servidor Publico do Estado de Sao Paulo, São Paulo
- France (2):
  - Centre Hospitalier Regional et Universitaire de Marseille, Service de Chirurgie Plastique Reparatrice et Esthetique, Marseille
  - Center Des Brules Hopital Cochin, Paris
- Germany (3):
  - Unfallkrankenhaus Berlin Burn Center, Berlin
  - BG - Unfallklinik Ludwigshafen, Ludwigshafen
  - Klinikum Mannheim Universtatsklinikum, Mannheim
- Soroka University Medical Center, Beersheba, Israel
- Italy (2):
  - Centro Grandi Ustionati, Cesena
  - Direttore U.O. Chirurgia Plastica e Centro Ustioni Ospedale Civico, Palermo
- Wojskowy Instytut Medyczny, Warsaw, Poland
- Emergency Clinic Hospital "Bagdazar-Arsenie", Bucharest, Romania
- Slovakia (2):
  - Center for Burns & Reconstructive Surgery, University Hopsital Bratislava, Bratislava
  - Clinic of Burns and Reconstructive Surgery Hospital Kosice, Kosice-Saca
- United Kingdom (2):
  - Queen Victoria Hospital, East Grinstead
  - The Burn Center Pinderfields Hospital, Wakefield

REFERENCES:
- [Background] Rosenberg L, Lapid O, Bogdanov-Berezovsky A, Glesinger R, Krieger Y, Silberstein E, Sagi A, Judkins K, Singer AJ. Safety and efficacy of a proteolytic enzyme for enzymatic burn debridement: a preliminary report. Burns. 2004 Dec;30(8):843-50. doi: 10.1016/j.burns.2004.04.010. PMID 15555800
- [Derived] Sinha S, Gabriel VA, Arora RK, Shin W, Scott J, Bharadia SK, Verly M, Rahmani WM, Nickerson DA, Fraulin FO, Chatterjee P, Ahuja RB, Biernaskie JA. Interventions for postburn pruritus. Cochrane Database Syst Rev. 2024 Jun 5;6(6):CD013468. doi: 10.1002/14651858.CD013468.pub2. PMID 38837237
- [Derived] Rosenberg L, Krieger Y, Bogdanov-Berezovski A, Silberstein E, Shoham Y, Singer AJ. A novel rapid and selective enzymatic debridement agent for burn wound management: a multi-center RCT. Burns. 2014 May;40(3):466-74. doi: 10.1016/j.burns.2013.08.013. Epub 2013 Sep 26. PMID 24074719